CLINICAL TRIAL: NCT04187807
Title: Efficacy of the Administration of Melatonin 5mg in the Prevention of Delirium in Older Adults Hospitalized in the Emergency Department
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Autonoma de San Luis Potosí (Other)
Responsible Party: Principal Investigator, Fátima Alondra Sánchez Martínez, Medical Doctor, Universidad Autonoma de San Luis Potosí
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UAutonomaSLP
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Delirium in Old Age
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: Parallel Assignament
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin 5mg (Experimental): Melatonin 5mg, every 24 hours for 14 days
  Interventions: Drug: Melatonin 5 mg
- Placebo (Placebo Comparator): Starch based placebo, every 24 hours for 14 days
  Interventions: Drug: Melatonin 5 mg

INTERVENTIONS:
Drug: Melatonin 5 mg — Placebo
  Other Names: Cronocaps

SUMMARY:
This study evaluates the efficacy of melatonin 5mg in the prevention of Delirium in the older adults in emergency department. Half of the participants will receive melatonin 5mg and the other half will use a starch-based placebo.

DETAILED DESCRIPTION:
Melatonia is useful for the treatment of sleep disorders due to the interruption of the circadian rhythm, secondary to alterations caused by the environment. The doses of 5 to 10mg oral or sublingual can improve the quality of the sleep-wake cycle and alertness in short-term use.

Mechanism of action of melatonin are:

1. Binding to membrane receptors: MT1 and MT2 coupled to G protein
2. - Union to nuclear receptors.
3. - Interaction with cytosolic proteins.
4. - Antioxidant of direct and indirect action.
5. - Interaction with mitochondria.

Melatonin circulates 80% bound to albumin and the rest in free form in plasma, 85-90% is metabolized by 6-hydroxymelatonin in the liver, which is then conjugated with sulfuric acid (70-80%) or glucuronic ( 5-3%), and is excreted in urine and feces.

Melatonin and its metabolites act as catalytic antioxidants to safeguard mitochondrial electron transfer reactions, therefore, increases the efficiency of energy metabolism. Melatonin synthesis decreases significantly as age progresses and changes in the circadian cycle have been associated with accelerated aging.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 60 who enter the emergency department with a stay in the ward for more than 8 hours and who will remain hospitalized for more than 48 hours due to admission pathology.
* Patients who agree to participate in the study by signing an informed consent (Signature by patient and / or family member).

Exclusion Criteria:

* Patients with a history of dementia or previous neurological diseases.
* Patients with a history of psychiatric disorder.
* Patients diagnosed with any type of liver disease.
* Warfarin treatment.
* Delirium data on admission to the emergency department.
* Patients under invasive mechanical ventilation and sedation.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Estimated)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Delirium | 14 days
  Diagnosis based Confusional Assessment Method Scale

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Gordillo, PhD, Study Director — Universidad Autonoma de San Luis Potosí; Fatima A Sánchez, Doctor of medicine, Principal Investigator — Universidad Autonoma de San Luis Potosí
Locations (1):
- Instituto Mexicano Del Seguro Social, San Luis Potosí City, Mexico

IPD SHARING:
Plan to Share IPD: No